CLINICAL TRIAL: NCT05643456
Title: Comparison Between The Results Of Operating Two Muscles And Operating Three Muscles For The Treatment Of Large Angle Exotropia
Brief Title: Surgery for Large Angle Exotropia Two Muscles Versus Three Muscles
Acronym: XT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, reham fawzy elsherbiny, assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIO
Record Dates: First submitted 2020-12-26; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Exotropia
MeSH Terms: conditions — Exotropia | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: 69 Patients with exotropia of (40-55) PD who are ≥ 5 years old. The 1st group will do two muscles surgery; bilateral lateral rectus recession. The 2nd group will do three muscles surgery; bilateral lateral rectus recession and unilateral medial rectus tucking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 :Two muscle surgery (Active Comparator): 30 patients will underwent two muscle surgery(bilateral lateral rectus muscle recession)
  Interventions: Procedure: surgery
- group 2:Three muscle surgery (Active Comparator): 39 patients underwent three muscle surgery(bilateral lateral rectus muscle recession with unilateral medial rectus muscle tucking)
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — 69 Patients with exotropia of (40-55) PD who are ≥ 5 years old. The 1st group 30 patients had two muscles surgery; bilateral lateral rectus recession.
  The 2nd group 39 patients had three muscles surgery; bilateral lateral rectus recession and unilateral medial rectus tucking.

SUMMARY:
Comparison Between The Results Of Two Muscles Surgery And Three Muscles Surgery For The Treatment Of Large Angle Exotropia

DETAILED DESCRIPTION:
Exotropia is classified as Primary which includes constant and intermittent exotropias. Secondary XT include Sensory and consecutive XT. Management for IXT consists of non-surgical and surgical treatment. There is some controversy regarding the optimal surgical method varying between bilateral lateral rectus recession (BLR), unilateral lateral rectus recession-medial rectus resection (RR) and bilateral medial rectus resection (BMR).

ELIGIBILITY:
Inclusion Criteria:

* Patients above age of 5 years with concomitant Exotropia of (40-55) PD of any type.

Exclusion Criteria:

1. Angle of deviation less than 40 PD or more than 55 PD.
2. History of previous surgery.
3. Inconcomitant exotropia.
4. Incomitance in any gaze.
5. Associated vertical deviation(oblique dysfunction,A or V pattern).
6. Patients with neurological deficit.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
alignment in the primary position | 1 week to 6 months
  measuring any misalignment by prism bar
palpebral fissure height | 1 week to 6 months
  measuring with millimeter
End gaze deficit | 1 week to 6 months
  measuring with prism bar

CONTACTS AND LOCATIONS:
Overall Officials: Lobna MH Khazbm, MD, Principal Investigator — Cairo University
Locations (1):
- Reham fawzy elsherbiny, Giza, Egypt